CLINICAL TRIAL: NCT03776201
Title: Merging Attentional Focus and Balance Training to Reduce Fall Risk in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Greensboro (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A18-0033; 1R15AG053866-01A1 (NIH)
Record Dates: First submitted 2018-11-16; First posted 2018-12-14 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2021-10

CONDITIONS: Accidental Fall

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internal Focus (Experimental): The internal focus group will receive 20 minutes of balance training 2 times per week. All training sessions will include a 5-minute walking warm-up, a 20-minute balance training program, and a 5-minute walking cool-down. The balance training will use a 30" wobble board with five bases ranging from 1" (easy) to 3" (very difficult). 20 trials of balance practice for 30-second intervals with 30-second breaks in between trials will be used every day. The Internal Focus group will be reminded to focus their attention internally via the prompt "keep your feet as level as possible" prior to each balance trial. To monitor whether the experimental groups are focusing as asked and to what extent, a compliance check that has been used in similar attentional focus literature will be used.
  Interventions: Other: Balance Training
- External Focus (Experimental): The external focus group will receive 20 minutes of balance training 2 times per week. All training sessions will include a 5-minute walking warm-up, a 20-minute balance training program, and a 5-minute walking cool-down. The balance training will use a 30" wobble board with five bases ranging from 1" (easy) to 3" (very difficult). 20 trials of balance practice for 30-second intervals with 30-second breaks in between trials will be used every day. The external focus group will be reminded to focus their attention externally via the prompt "please keep the board as level as possible" prior to each balance trial. To monitor whether the experimental groups are focusing as asked and to what extent, a compliance check that has been used in similar attentional focus literature will be used.
  Interventions: Other: Balance Training
- Control (No Intervention): The control group will not receive any balance training

INTERVENTIONS:
Other: Balance Training — We expect that a balance training intervention that utilizes an external focus of attention will lead to the adoption of balance strategies that are protective against falls. The mechanism for this behavioral change will be identified using a Dynamical Systems Theory framework (i.e., entropy) to quantify postural sway characteristics before, during and after the training. We will determine whether the balance intervention utilizing an external focus of attention will lead to positive benefits through the three specific aims.
  Arms: External Focus; Internal Focus

SUMMARY:
Approximately 15 million older adults fall every year in the United States and fall prevention programs have only been moderately successful in arresting fall rates. This proposal uses motor learning principles derived from the attentional focus literature to determine whether training someone where to focus their attention during a balance task enhances balance control and reduces fall risk. Older adults (N=90) who are classified as fallers (one or more falls in the past 12 months) will be recruited. A series of balance control, clinical metrics of fall risk, and patient-reported outcomes will be assessed prior, during, and after a 12-week intervention to examine changes in performance and fall risk. The 12-week intervention will emphasize directing the participants' attention either internally or externally during a series of balance tasks. Empirical evidence and our preliminary data leads us to hypothesize that an external focus of attention training will positively influence balance control. This will be the first study to will examine balance control changes over 12-week balance intervention using an attentional focus paradigm and we will relate the balance control changes to clinical metrics that indicate fall risk and patient-reported outcomes. Further, our proposal includes a novel model of entropy in postural sway, a metric that has been proposed to relate to balance ability, to help explain the hypothesized enhancement in balance. Thus, this proposal will merge motor learning principles with a 12-week balance intervention to determine if fall risk is reduced in older adults. Specific Aim 1 compares balance performance within each trial/session throughout the 12 weeks of balance training to evaluate whether the attentional focus groups (external vs. internal) differ in their motor learning trajectory with respect to the balance task. Specific Aim 2 compares the motor ability outcome measures that relate to fall-risk between the groups (external focus, internal focus, or control) before, during, and after the 12-week balance intervention. Specific Aim 3 compares the patient-reported outcome measures of fear of falling, functional health and well-being, and fear of injury from movement between the groups (external focus, internal focus, or control) before, during, and after the 12-week balance intervention.

DETAILED DESCRIPTION:
Falls due to poor balance are common and costly in older adults. Unfortunately, traditional balance interventions show mixed results in reducing falls. Balance is controlled by a complex system that depends on a host of cognitive functions, including attention. While attention has different meanings in different research areas, this proposal will examine attention defined as a performer's conscious perception of information for a task, which can be focused internally or externally. An internal focus of attention is directed at the performer's own body movements, while an external focus is directed at the effects a particular movement has on the environment. Fall prevention interventions typically emphasize an internal focus of attention. However, mounting evidence from laboratory settings indicates that an external focus of attention improves balance control. For example, participants in one study were asked to balance on a stabilometer, which is an unstable device that swings forward or backward when someone is out of balance. Participants were asked to focus on keeping their feet level (i.e., an internal focus) or keeping the surface of the stabilometer level (i.e., an external focus). When the participants adopted an external focus, their balance was enhanced. That is, they had fewer deviations from their starting position (i.e., less variability in their motion). Follow-up research also showed that participants were able to respond faster to their change in body position during a balance task when they adopted an external focus. Both of these characteristics would be beneficial for an older adult population with a history of falls.

The theoretical explanation of these findings is the constrained-action hypothesis, which suggests that an internal focus of attention constrains the system in a way that does not allow it to find an optimal solution. For example, instructions that ask a participant to focus internally by keeping their feet level may constrain other parts of the body and actually diminish balance control. In contrast, instructions that ask a participant to focus externally by keeping a balance apparatus level allow the body to find the optimal way to perform the task. This small change in instruction has been repeatedly shown to significantly enhance performance. Thus, emphasizing an external focus of attention may be critical to the optimization of strategies designed to improve balance and reduce fall risk in older adults. This approach does not require a re-tooling of all clinical practice, just a modification of current delivery, making the cost-benefit ratio of the approach appealing to clinical practitioners and administrators. The goal of this proposed study, therefore, is to extend this line of research to determine the efficacy of using an external focus of attention to enhance balance control and decrease fall risk in older adults.

To show proof-of-concept, we conducted 2 preliminary studies. The 1st preliminary study showed that older adults who adopted an external focus of attention during a balance task had greater postural control complexity, which is typically interpreted as a more adaptable and less fall-prone behavior. The 2nd preliminary study showed that an external focus of attention increases the time-in-balance for older adults standing on a wobble board. By altering the attentional focus, our data show that the external focus instructions lead to more stable postural control. This is consistent with the plethora of literature showing the positive effect of adopting an external focus of attention on motor control performance. These preliminary results give us confidence that a 12-week balance intervention that emphasizes an external focus of attention will be superior to a similar intervention that utilizes an internal focus of attention (i.e., what is used in traditional balance interventions). Balance control, clinical metrics of fall risk, and patient-reported outcomes of functional ability will be recorded before, during, and after a 12 week balance training intervention in a cohort of 90 older adults with a history of falls. There are three specific aims for this proposal:

SPECIFIC AIM 1: Compare balance performance within each trial/session to evaluate whether the attentional focus groups (external vs. internal) differ in their motor learning trajectory with respect to the balance task.

Hypothesis 1: The external focus group will exhibit a faster rate of motor learning toward stable balance.

SPECIFIC AIM 2: Compare the motor ability outcome measures that relate to fall-risk between the groups (external focus, internal focus, or control) before, during, and after the 12 week balance intervention.

Hypothesis 2a: The external focus group will exhibit a greater reduction in fall-risk during mid- and post-testing relative to the internal focus and control groups.

Hypothesis 2b: Sensory information (vision, vestibular, and somatosensory scores) and attention will be related to fall risk, but mediated through entropy of postural sway.

SPECIFIC AIM 3: Compare the patient-reported outcome measures of fear of falling, functional health and well-being, and fear of injury from movement between the groups (external focus, internal focus, or control) before, during, and after the 12 week balance intervention.

Hypothesis 3: The external focus group will have a significantly lower fear of falling, enhanced functional health and well-being, and lower fear of injury from movement during mid- and post-testing relative to the internal focus and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Older adults (N=90) who are classified as fallers (≥ 1 fall in the last 12 months) will be recruited

Exclusion Criteria:

* • Younger than 65 or older than 90 years old

  * Failure to receive medical clearance from their physician to participate in the study and confirming that their patient has fallen at least once within the last 12 months
  * Inability to walk independently for at least 10 consecutive minutes
  * Score in the "impaired" range on the Mini-Mental State Examination, adjusted for age and education level [60].
  * A diagnosis of a neurological disorder that requires medication
  * A visual impairment of 20/70 or worse
  * A body mass index of ≥ 30
  * Any acute medical problems, including musculoskeletal based impairments, that lead to pain or discomfort during standing or walking

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the BTracks measurement | Weeks 0, 6, 12, 13, 16, 20
  The average measurement of the center of pressure displacement during three 20-second trials with eyes closed
Change in the Functional Gait Assessment | Weeks 0, 6, 12, 13, 16, 20
  Assesses postural stability during walking tasks
Change in the Timed Up and Go | Weeks 0, 6, 12, 13, 16, 20
  Assesses a person's mobility and requires both static and dynamic balance.
Change in the Berg Balance Test | Weeks 0, 6, 12, 13, 16, 20
  Assesses the static standing balance and subsequent fall risk
Change in the Activities Balance Confidence Scale short version | Weeks 0, 6, 12, 13, 16, 20
  Assesses the Fear of Falling. The scale is from 0-100% for the overall scores. The scores from each of the 16 questions (which range from 0-100%) are summed and then divided by 16 to get the overall score. A high score equates to greater function.
Change in the Short Form 36 | Weeks 0, 6, 12, 13, 16, 20
  The SF-36 is a measure of health status. Scoring the RAND 36-Item Health Survey is a two-step process. First, precoded numeric values are recoded per the scoring key given. Note that all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores. Items that are left blank (missing data) are not taken into account when calculating the scale scores. Hence, scale scores represent the average for all items in the scale that the respondent answered.
Change in the Tampa Scale of Kinesiophobia | Weeks 0, 6, 12, 13, 16, 20
  The Tampa Scale of Kinesiophobia measures the fear of injury from movement on a range of 17-68, with high scores indicating high fear of movement related injury. A cutoff score of 37 indicates increased fear of injury from movement

SECONDARY OUTCOMES:
Change in the XSens - Time in Balance - Anterior Posterior | Assessed at the end of each training session, which is provided 2 times per week for 12 weeks. Thus, this variable is assessed a total of 24 times. After the 24 sessions, the timeframe is complete for this outcome.
  Duration in which the wobble board is +/- 3 deg of a neutral position (0 deg) in the anterior-posterior direction for 30 seconds
Change in the XSens - Time in Balance - Medial Lateral | Assessed at the end of each training session, which is provided 2 times per week for 12 weeks. Thus, this variable is assessed a total of 24 times. After the 24 sessions, the timeframe is complete for this outcome.
  Duration in which the wobble board is +/- 3 deg of a neutral position (0 deg) in the medial-lateral direction for 30 seconds
Change in the XSens - Mean Power Frequency - Anterior Posterior | Assessed at the end of each training session, which is provided 2 times per week for 12 weeks. Thus, this variable is assessed a total of 24 times. After the 24 sessions, the timeframe is complete for this outcome.
  Mean power frequency of the wobble board in the anterior-posterior direction for 30 seconds
Change in the XSens - Mean Power Frequency - Medial Lateral | Assessed at the end of each training session, which is provided 2 times per week for 12 weeks. Thus, this variable is assessed a total of 24 times. After the 24 sessions, the timeframe is complete for this outcome.
  Mean power frequency of the wobble board in the medial-lateral direction for 30 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Louisa D Raisbeck, PhD, Principal Investigator — University of North Carolina, Greensboro
Locations (1):
- UNCG Motor Behavior, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No